CLINICAL TRIAL: NCT06803719
Title: Public Awareness, Trust, and Risk Perception Toward Robotic Surgery, Telesurgery and Telemedicine
Brief Title: Public Perceptions Toward Robotic Surgery, Telesurgery and Telemedicine
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Ling Zhan, Principal Investigator, Shanghai 6th People's Hospital
Other Study IDs: 2025-KY-507(K)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Robotic Surgery; Telemedicine
Keywords: Public perception; Telemedicine adoption; Surgical training; Surgical decision-making
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Public group: The general public sample included residents of mainland China aged 18 and older who were able to understand and complete the questionnaire, regardless of gender, region, or occupation. The aim was to assess the general public's awareness, risk perception, trust, and acceptance of robotic surgery and remote surgery.
  Interventions: Other: Survey Questionnaire
- Physician group: The clinical physician sample included practicing physicians from surgical specialties (such as general surgery, urology, gynecology, thoracic surgery, thyroid surgery, etc.), including residents, attending physicians, and chief/deputy chief physicians of different seniority levels. This group of physicians was used to assess healthcare professionals' awareness, experience, perceived risks, expectations for future applications of robotic and remote surgery, as well as their views on training needs, feasibility, and barriers to training.
  Interventions: Other: Survey Questionnaire

INTERVENTIONS:
Other: Survey Questionnaire — Anonymous online questionnaire assessing public and physician perceptions of robotic surgery, telesurgery and telemedicine

SUMMARY:
This study aims to systematically assess the public's and clinicians' levels of awareness, attitudes, risk perception, acceptance, and potential concerns regarding robotic surgery and telesurgery. It also analyzes the key factors influencing their attitudes and explores the needs of physicians regarding training systems for robotic and telesurgery, as well as the factors affecting their preparedness.

DETAILED DESCRIPTION:
Public level:

* Level of awareness and understanding of robotic and remote surgery (e.g., understanding of operating procedures, the doctor's role, and potential risks).
* Perceptions and concerns regarding the safety, reliability, cybersecurity risks, and equipment malfunctions of the technology.
* Trust and acceptance of the technology, and factors that may influence attitudes (e.g., education level, past medical experiences, access to medical resources).
* Overall expectations and concerns regarding hospitals performing such surgeries.

Healthcare practitioners level:

* Knowledge level, attitudes, and acceptance of robotic and remote surgery.
* Views on the learning curve, surgical safety, equipment accessibility, collaborative processes, and potential obstacles.
* Understanding and actual needs regarding training systems for robotic and remote surgery, including simulator training, mentorship programs, skill evaluation methods, and the transfer of laparoscopic skills to robotic skills.

ELIGIBILITY:
Inclusion Criteria:

* Chinese citizens aged 18 years or older
* Able to understand and complete the questionnaire
* Voluntarily participating in this study and providing informed consent

Exclusion Criteria:

* Aged below 18 years
* Unable to understand the questionnaire or unable to complete the questionnaire independently
* Those who submit the questionnaire repeatedly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The general public sample included residents of mainland China aged 18 and older who were able to understand and complete the questionnaire, regardless of gender, region, or occupation. The aim was to assess the general public's awareness, risk perception, trust, and acceptance of robotic surgery and remote surgery. The clinical physician sample included practicing physicians from surgical specialties (such as general surgery, urology, gynecology, thoracic surgery, thyroid surgery, etc.), including residents, attending physicians, and chief/deputy chief physicians of different seniority levels.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Public acceptance of robotic surgery | Baseline
  The level of acceptance toward robotic surgery among the general public, measured using a 5-point Likert scale assessing willingness to receive robotic-assisted procedures under hypothetical clinical scenarios. Higher scores indicate greater acceptance.
Public acceptance of telesurgery and telemedicine | Baseline
  The degree of acceptance of telesurgery among the general public, assessed via a validated questionnaire evaluating willingness to undergo remote surgery, perceived safety, and perceived reliability of network-based surgical systems.
Public perceived risk of robotic and telesurgery | Baseline
  Perceived risk associated with robotic surgery and telesurgery, including concerns about device malfunction, network failure, surgical autonomy, and responsibility attribution, assessed using a multi-item Likert scale. Higher scores indicate higher perceived risk.
Physicians' training needs score (assessed by self-designed questionnaire) | Baseline
  This measure assesses physicians' perceived training needs regarding required skills (e.g., simulation, console operation) and preferred modalities (e.g., online courses, wet labs). Participants rate items on a 5-point Likert scale (1=Not needed, 5=Highly needed).

CONTACTS AND LOCATIONS:
Overall Officials: Ling Zhan, Dr, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data are available on request due to privacy or other restrictions. The data that support the findings of this study are available on request from Ling Zhan. The data are not publicly available due to them containing information that could compromise research participant privacy.